CLINICAL TRIAL: NCT03551704
Title: Smoking Cessation Treatment for Substance Use Dependents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Roberto Secades-Villa, PhD, Professor, PhD, University of Oviedo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSSSI-2017-2017I036
Record Dates: First submitted 2018-05-09; First posted 2018-06-11 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Tobacco Use Disorder
Keywords: Smoking; Substance addiction; Cocaine; Alcohol; Behavioral treatment
MeSH Terms: conditions — Tobacco Use Disorder; Smoking; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to each of the two treatment conditions in accordance with a computer-generated randomization list. The treatment conditions will be actively running in parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT + EFT (Active Comparator): The CBT treatment will be implemented in 8-week group-based sessions (maximum 4 patients). Sessions will be carried out once a week over an 8-week period, with quit date occurring at fifth session. Patients will be asked to gradually reduce their nicotine intake (i.e., 25% each week). CBT components include: psychoeducation, self-monitoring, physiological feedback, training in stimulus control and strategies for controlling negative discomfort, and relapse prevention strategies.
  As part of the EFT, participants will be asked to select future smoking-related events that would occur within the following time periods: 2 weeks, 1, and 6 months. They will be instructed to generate personal audio recordings that will be used to help them think about future decision-making choices.
  Interventions: Behavioral: CBT + EFT
- CBT + EFT + CM (Experimental): This intervention includes the abovementioned treatment components and a CM procedure reinforcing abstinence. This arm will consist on delivering CBT and EFT and providing patients incentives to promote and reinforce abstinence contingent on biochemical verification. The schedule will incorporate an increasing magnitude of reinforcement.
  Interventions: Behavioral: CBT + EFT + CM

INTERVENTIONS:
Behavioral: CBT + EFT — The CBT treatment will be implemented in 8-week group-based sessions (maximum 4 patients). Sessions will be carried out once a week over an 8-week period, with quit date occurring at fifth session. Patients will be asked to gradually reduce their nicotine intake (i.e., 25% each week). CBT components include: psychoeducation, self-monitoring, physiological feedback, training in stimulus control and strategies for controlling negative discomfort, and relapse prevention strategies.
  As part of the EFT, participants will be asked to select future smoking-related events that would occur within the following time periods: 2 weeks, 1, and 6 months. They will be instructed to generate personal audio recordings that will be used to help them think about future decision-making choices.
  Arms: CBT + EFT
Behavioral: CBT + EFT + CM — This intervention includes the abovementioned treatment components and a CM procedure reinforcing abstinence. This arm will consist on delivering CBT and EFT and providing patients incentives to promote and reinforce abstinence contingent on abstinence. The schedule will incorporate an increasing magnitude of reinforcement.
  Arms: CBT + EFT + CM

SUMMARY:
The present research project aims to develop an innovative and empirically validated intervention protocol for smoking cessation among patients with substance use disorders (SUDs). For this purpose, two smoking cessation treatments tailored for SUDs will be assessed. Participants will be assigned to one of the following treatment conditions: 1) Cognitive-behavioral treatment for smoking cessation (CBT) + Episodic Future Thinking (EFT); 2) The same treatment alongside Contingency Management (CM) for shaping abstinence.

The main goals are:

1. To analyze the feasibility (e.g., acceptability, compliance) of implementing the abovementioned protocol treatments to a community setting.
2. To assess abstinence rates in each treatment condition at short and long-term follow-ups: post-treatment, one, two, three, six and twelve months after post-treatment.
3. To assess the effects of smoking abstinence on other substance use.
4. To analyze the moderating effect of individual variables over treatment outcomes: sociodemographic characteristics, drug demand, severity of nicotine dependence and SUD, severity of depressive symptomatology and impulsivity.

DETAILED DESCRIPTION:
Cigarette smoking continues to have a startling adverse impact on public health, leading to more than 5 million premature deaths annually worldwide. Smoking rates are disproportionately high among the population suffering from substance use disorders (SUDs) (e.g., alcohol or cocaine). In this regard, smokers with comorbid SUD are more likely to smoke heavily and meet criteria for high nicotine dependence. As they experience more difficulty in quitting smoking than their non-SUDs counterparts, they present lower rates of abstinence.

In recent years there has been a great interest in developing effective strategies to promote abstinence in smokers with SUDs. In particular, a proliferation on CM treatments for smokers with SUDs has been recently produced. There is promising evidence for the positive effect of CM treatments upon both quitting smoking and both legal and illegal abuse drugs. On the other hand, CM has shown promising results in promoting both retention and nicotine abstinence among comorbid and non-comorbid smokers. Nevertheless, there is a lack of research exploring the effectiveness of CM on smokers with SUDs.

The primary aim of this clinical trial is to yield data on the effectiveness of CM for smoking cessation in smokers with SUDs. To address this issue, both CBT for smoking cessation plus EFT, and the same treatment alongside CM for shaping abstinence will be assessed. Participants will be randomly assigned to one of the following treatment conditions: 1) CBT+EFT; 2) CBT+EFT+ CM.

In view to assure adequate power for achieving statistical significance, investigators carried out a priori power analysis by using the G*Power 3.1. An estimated sample size of 120 participants would detect a medium effect size (Cohen's d = 0.3, with power (1-β) set at 0.97 and α = 05).

The primary analyses derived from this clinical trial will be conducted using Statistical Package for the Social Science (SPSS) version 24 for Windows. A set of descriptive and frequency analyses will be carried out with regard to participants' characteristics. Comparisons between treatment groups in both baseline characteristics and treatment outcomes will be conducted using a set of chi-square tests for categorical variables and t-tests (two-tailed) for continuous variables.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 18 or over.
* Having smoked 10 or more cigarettes/day within the last year.
* Meeting the diagnostic criteria for nicotine dependence according to the Diagnostic and Statistical Manual of Mental Disorders-5th ed. (American Psychiatric Association 2013).
* Undergoing outpatient cocaine or alcohol treatment.

Exclusion Criteria:

* Not being able to attend the entire treatment.
* Being currently receiving other psychological/pharmacological treatment for smoking cessation.
* Being diagnosed with a current severe psychiatric disorder (i.e., schizophrenia,bipolar disorder).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in Smoking Abstinence | End-of-treatment (8-week), 1, 2, 3, 6 and 12 month follow-up
  Abstinence is defined as achieving a period of at least 24 hours of abstinence (end-of-treatment) or not smoking since the prior last 7 days. Abstinence is assessed by means of carbon monoxide (CO) and cotinine samples.
Changes in Continuous abstinence | 1, 2, 3, 6 and 12 month follow-up since the treatment completion
  Abstinence is defined as no smoking (not even a puff) since the participant´s quit day. Abstinence is assessed by means of carbon monoxide (CO) and cotinine samples.

SECONDARY OUTCOMES:
Changes in Other Substance Abstinence | End-of-treatment (8-week), 1, 2, 3, 6 and 12 month follow-up since the treatment completion
  7-day point-prevalence. Self-reported abstinence will be confirmed by urinalyses and breath alcohol samples.
Changes in Drug demand | Intake (baseline), end-of-treatment (8-week),1,2,3,6 and 12 months follow-up since treatment completion
  Alcohol and tobacco demand will be assessed by using the Alcohol and Tobacco Purchase Task. These tasks allow to capture changes in the relative reinforcing efficacy of different drugs through the course of treatment. From this tasks, five demand indices are derived. Specifically, we will compute the indices that follow:
  Breakpoint: The first price at which consumption is zero
  Omax: maximum expenditure for cigarettes
  Pmax: price at which expenditure is maximized
  Intensity: consumption at the lowest price
  Elasticity: sensitivity of cigarette consumption to increases in costs
Changes in Health-Related Quality of Life | Intake (baseline), end-of-treatment (8-week),1,2,3,6 and 12 months follow-up since treatment completion
  This variable will be assessed by using the EuroQol-5D (EQ-5D). It essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions.
Changes in Depression | Intake (baseline), end-of-treatment (8-week),1,2,3,6 and 12 months follow-up since treatment completion
  Depression will be assessed using the Beck's Depression Inventory- Second Edition (BDI-II). Scores are examined as a continuous scale. None/minimal depression is defined as scoring below the clinical screening BDI cutoff of mild depression (<14). Depression diagnosis is assessed in those individuals scoring 14 or more on the BDI-II by means of the Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders-Clinical Version (SCID-I/CV).
Changes in Impulsivity | Intake (baseline), end-of-treatment (8-week),1,2,3,6 and 12 months follow-up since treatment completion
  Impulsivity levels will be assessed by means of the delay discounting task. Participants will complete a computerized version of this task and will be presented with several choices. An adjusting-amount procedure will be used (Holt, Green, & Myerson, 2012). The delay values used are one day, one week, one month, six months, one year, five years, and 25 years. Delay discounting is calculated using logk and the area under the curve (AUC).
Cost Analysis | End of the project when all participant´s data are collected. Data expected: three years after the study onset.
  The Drug Abuse Treatment Cost Analysis Program (DATCAP) is a cost data collection instrument and interview guide designed to be used in a variety of medical treatment and social service settings.
  The instrument is intended to collect and organize detailed information on resources used in service delivery and their associated dollar cost. Resource categories include personnel, supplies and materials, contracted services, buildings and facilities, equipment, and miscellaneous items.
  The Drug Abuse Treatment Cost Analysis Program (DATCAP) is a cost data collection instrument and interview guide designed to be used in a variety of medical treatment and social service settings.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Secades-Villa, PhD, Principal Investigator — University of Oviedo
Locations (1):
- Clinical Unit of Addictive Behaviors, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Secades-Villa R, Gonzalez-Roz A, Garcia-Perez A, Becona E. Psychological, pharmacological, and combined smoking cessation interventions for smokers with current depression: A systematic review and meta-analysis. PLoS One. 2017 Dec 5;12(12):e0188849. doi: 10.1371/journal.pone.0188849. eCollection 2017. PMID 29206852
- [Result] McKelvey K, Thrul J, Ramo D. Impact of quitting smoking and smoking cessation treatment on substance use outcomes: An updated and narrative review. Addict Behav. 2017 Feb;65:161-170. doi: 10.1016/j.addbeh.2016.10.012. Epub 2016 Oct 27. PMID 27816663
- [Result] Secades-Villa R, Vallejo-Seco G, Garcia-Rodriguez O, Lopez-Nunez C, Weidberg S, Gonzalez-Roz A. Contingency management for cigarette smokers with depressive symptoms. Exp Clin Psychopharmacol. 2015 Oct;23(5):351-60. doi: 10.1037/pha0000044. Epub 2015 Aug 17. PMID 26280589
- [Result] Weidberg S, Vallejo-Seco G, Gonzalez-Roz A, Garcia-Perez A, Secades-Villa R. In-treatment cigarette demand among treatment-seeking smokers with depressive symptoms. Addict Behav. 2018 Jul;82:35-43. doi: 10.1016/j.addbeh.2018.02.022. Epub 2018 Feb 16. PMID 29482033
- [Result] Cooney JL, Cooper S, Grant C, Sevarino K, Krishnan-Sarin S, Gutierrez IA, Cooney NL. A Randomized Trial of Contingency Management for Smoking Cessation During Intensive Outpatient Alcohol Treatment. J Subst Abuse Treat. 2017 Jan;72:89-96. doi: 10.1016/j.jsat.2016.07.002. Epub 2016 Jul 15. PMID 27542442